CLINICAL TRIAL: NCT03272841
Title: TransplantLines: the Transplantation Biobank
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof. dr. S.J.L. Bakker, MD, PhD, Internist-nephrologist, University Medical Center Groningen
Other Study IDs: TXLINES01
Record Dates: First submitted 2017-09-02; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Solid Organ Tranplant Recipients, 18+ Years

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — 1x serum
  1x EDTA
  1x Lithium-heparine
  1x Citrate
  1x PAXgene Faeces, hair and nails
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Transplant recipients: Renal, heart, lung, liver, small bowel, pancreas or combined transplant recipients

SUMMARY:
TransplantLines is an observational cohort study in all solid transplant recipients, i.e. kidney, heart, lung, liver, small bowel and pancreas. In this study we will gather questionnaires about topics affecting transplant recipients, e.g. QoL, work and physical capacity. Moreover, we will collect multiple urine and blood samples for analysis. Additionally, we will store hair, nails and faeces from the transplant recipients. Next to this, we will perform physical capacity tests and cognitive tests.

DETAILED DESCRIPTION:
The last decades, the acute period after transplantation has markedly improved due to improved tissue-matching techniques and better immunosuppressive drugs. However, nowadays the major aim after transplantation is the long-term patient and graft survival which are still poor, where half of the RTR looses their graft after 10 years. With TransplantLines we are setting up an extensive biobank to improve the long-term survival after transplantation. Moreover, we are one of the few studies to collect across transplant specialities. Like mentioned in the brief summary, extensive questionnaires will be send to participants prior to the visit containing multiple questionnaires (e.g. SF-36, WHODAS, PQ-SGA etc.). During the visit, we will collect multiple blood samples who will be taken during the regularly visit to the clinician. Moreover, two tubes from 24-hour urine collection will be collected, faeces, hair and nails will be stored. Finally, physical tests and cognitive tests will be performed with the participants (e.g. 2-min walking test, 4m walking test, timed-up-and-go test etc.).

ELIGIBILITY:
Inclusion Criteria:

* Solid organ transplant recipients

Exclusion Criteria:

* Age younger than 18 years old
* Cognitive dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All solid organ transplantation patients
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-06; Primary Completion 2020-09 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Graft failure / mortality | Untill 2020
  Development of graft failure or mortality in the transplant recipients

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Zorgdrager M, Liu Y, Hong J, Ghildayal N, Swaab TDA, Bakker SJL, Viddeleer AR, Orandi BJ, Shafaat O, Weiss CR, Segev D, McAdams-DeMarco M, Pol RA. Association of Myosteatosis and of Graft Loss after Kidney Transplantation: An International Observational Study. Clin J Am Soc Nephrol. 2026 Jan 1;21(1):118-129. doi: 10.2215/CJN.0000000862. Epub 2025 Oct 15. No abstract available. PMID 41091560
- [Derived] Yepes-Calderon M, Martin Del Campo Sanchez F, Kremer D, Knobbe TJ, Gomes Neto AW, Connelley MA, Dullaart RPF, Corpeleijn E, de Borst MH, Bakker SJL; TransplantLines Investigators. Plasma trimethylamine N-oxide concentration and all-cause mortality in kidney transplant recipients. Nephrol Dial Transplant. 2025 Sep 29;40(10):1931-1940. doi: 10.1093/ndt/gfaf071. PMID 40275497
- [Derived] Westenberg LB, Pol RA, van der Weijden J, de Borst MH, Bakker SJL, van Londen M; on behalf of the Transplant Lines Investigators. Central Body Fat Distribution and Kidney Function after Living Kidney Donation. Clin J Am Soc Nephrol. 2024 Apr 1;19(4):503-513. doi: 10.2215/CJN.0000000000000403. Epub 2024 Jan 8. PMID 38190119
- [Derived] Riemersma NL, Kremer D, Knobbe TJ, Gan CT, Nolte S, Gomes-Neto AW, Blokzijl H, de Meijer VE, Damman K, Eisenga MF, Drost G, Elting JWJ, Touw DJ, Berger SP, Bakker SJL, van der Stouwe AMM; Transplantlines Investigators. Tremor, Daily Functioning, and Health-Related Quality of Life in Solid Organ Transplant Recipients. Transpl Int. 2023 Mar 16;36:10951. doi: 10.3389/ti.2023.10951. eCollection 2023. PMID 37008718
- [Derived] van Vliet IMY, Post A, Kremer D, Boslooper-Meulenbelt K, van der Veen Y, de Jong MFC, Pol RA; TransplantLines Investigators; Jager-Wittenaar H, Navis GJ, Bakker SJL. Muscle mass, muscle strength and mortality in kidney transplant recipients: results of the TransplantLines Biobank and Cohort Study. J Cachexia Sarcopenia Muscle. 2022 Dec;13(6):2932-2943. doi: 10.1002/jcsm.13070. Epub 2022 Oct 6. PMID 36891995
- [Derived] Knobbe TJ, Kremer D, Abma FI, Annema C, Berger SP, Navis GJ, van der Mei SF, Bultmann U, Visser A, Bakker SJL; TransplantLines Investigators. Employment Status and Work Functioning among Kidney Transplant Recipients. Clin J Am Soc Nephrol. 2022 Oct;17(10):1506-1514. doi: 10.2215/CJN.05560522. PMID 36162849
- [Derived] Vinke JSJ, Wouters HJCM, Stam SP, Douwes RM, Post A, Gomes-Neto AW, van der Klauw MM, Berger SP, Bakker SJL; TransplantLines Investigators; De Borst MH, Eisenga MF. Decreased haemoglobin levels are associated with lower muscle mass and strength in kidney transplant recipients. J Cachexia Sarcopenia Muscle. 2022 Aug;13(4):2044-2053. doi: 10.1002/jcsm.12999. Epub 2022 Jun 3. PMID 35666066
- [Derived] Sotomayor CG, Giubergia F, Groothof D, Ferreccio C, Nolte IM, Navis GJ, Gomes-Neto AW, Kremer D, Knobbe TJ, Eisenga MF, Rodrigo R, Touw DJ, Bakker SJL; TransplantLines Investigators. Plasma Lead Concentration and Risk of Late Kidney Allograft Failure: Findings From the TransplantLines Biobank and Cohort Studies. Am J Kidney Dis. 2022 Jul;80(1):87-97.e1. doi: 10.1053/j.ajkd.2021.10.009. Epub 2021 Dec 4. PMID 34871698
- [Derived] Shahabeddin Parizi A, Vermeulen KM, Gomes-Neto AW, van der Bij W, Blokzijl H, Buskens E, Bakker SJ, Krabbe PF. Using a novel concept to measure outcomes in solid organ recipients provided promising results. J Clin Epidemiol. 2021 Nov;139:96-106. doi: 10.1016/j.jclinepi.2021.07.005. Epub 2021 Jul 14. PMID 34273526
- [Derived] Douwes RM, Swarte JC, Post A, Annema C, Harmsen HJM, Bakker SJL. Discrepancy between self-perceived mycophenolic acid-associated diarrhea and stool water content after kidney transplantation. Clin Transplant. 2021 Jul;35(7):e14321. doi: 10.1111/ctr.14321. Epub 2021 May 2. PMID 33882147
- [Derived] Nolte S, van Londen M, Elting JWJ, de Greef BTA, Kuks JBM, Faber CG, Nolte IM, Groen RJM, Bakker SJL, Groothof D, Lesman-Leegte I, Berger SP, Drost G. Vibration threshold in non-diabetic subjects. PLoS One. 2020 Oct 7;15(10):e0237733. doi: 10.1371/journal.pone.0237733. eCollection 2020. PMID 33027294
- [Derived] Hijmans RS, van Londen M, Sarpong KA, Bakker SJL, Navis GJ, Storteboom TTR, de Jong WHA, Pol RA, van den Born J. Dermal tissue remodeling and non-osmotic sodium storage in kidney patients. J Transl Med. 2019 Mar 18;17(1):88. doi: 10.1186/s12967-019-1815-5. PMID 30885222
- [Derived] Hessels AC, van der Hoeven JH, Sanders JSF, Brouwer E, Rutgers A, Stegeman CA. Leg muscle strength is reduced and is associated with physical quality of life in Antineutrophil cytoplasmic antibody-associated vasculitis. PLoS One. 2019 Feb 4;14(2):e0211895. doi: 10.1371/journal.pone.0211895. eCollection 2019. PMID 30716132
- [Derived] Eisenga MF, Gomes-Neto AW, van Londen M, Ziengs AL, Douwes RM, Stam SP, Oste MCJ, Knobbe TJ, Hessels NR, Buunk AM, Annema C, Siebelink MJ, Racz E, Spikman JM, Bodewes FAJA, Pol RA, Berger SP, Drost G, Porte RJ, Leuvenink HGD, Damman K, Verschuuren EAM, de Meijer VE, Blokzijl H, Bakker SJL. Rationale and design of TransplantLines: a prospective cohort study and biobank of solid organ transplant recipients. BMJ Open. 2018 Dec 31;8(12):e024502. doi: 10.1136/bmjopen-2018-024502. PMID 30598488